CLINICAL TRIAL: NCT01153763
Title: A Phase II (BRF113710) Single-arm, Open-label Study of GSK2118436 in BRAF Mutant Metastatic Melanoma
Brief Title: A Study of GSK2118436 in BRAF Mutant Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113710
Record Dates: First submitted 2010-05-27; First posted 2010-06-30 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-07

CONDITIONS: Melanoma
Keywords: Metastatic melanoma; BRAF mutant; Melanoma; BRAF mutant metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Other): Subjects will receive 150 mg of GSK2118436 twice daily and continue on treatment until disease progression, death, or unacceptable adverse event.
  Interventions: Drug: GSK2118436

INTERVENTIONS:
Drug: GSK2118436 — Subjects will receive 150 mg of GSK2118436 twice daily and continue on treatment until disease progression, death, or unacceptable adverse event.

SUMMARY:
BRF113710 is a Phase II, single-arm, open-label study to assess the efficacy, safety, and tolerability of GSK2118436 administered twice daily as a single agent in subjects with BRAF mutant metastatic melanoma. Subjects will receive 150 mg of GSK2118436 twice daily and continue on treatment until disease progression, death, or unacceptable adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must have histologically confirmed cutaneous metastatic melanoma (Stage IV) that is BRAF mutation-positive (V600 E/K) as determined via central testing with a BRAF mutation assay.
* Is treatment naive or has received prior treatment for metastatic melanoma.
* Must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Women of child-bearing potential must have a negative pregnancy test within 14 days prior to the first dose of study treatment.
* Women with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 4 weeks after the last dose of study medication.
* Men with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 16 weeks after the last dose of study medication.
* Must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate organ function.

Exclusion Criteria:

* Previous treatment with a BRAF or MEK inhibitor.
* Cancer therapy (chemotherapy with delayed toxicity, radiation therapy, immunotherapy, biologic therapy, or major surgery) within the last 3 weeks; chemotherapy regimens without delayed toxicity within the last 2 weeks; or use of any investigational anti-cancer or other drug within 28 days or 5 half-lives, whichever is longer, preceding the first dose of GSK2118436.
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection.
* History or evidence of brain metastases on MRI or head CT if MRI is not able to be performed.
* History of other malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Certain cardiac abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-08-09; Primary Completion 2011-07-01 (Actual); Study Completion 2016-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (5):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
- Australia (3):
  - GSK Investigational Site, Newcastle, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Nedlands, Western Australia
- France (7):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villejuif
- Germany (4):
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Italy (3):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Padua, Veneto

REFERENCES:
- [Background] Ascierto PA, Minor D, Ribas A, Lebbe C, O'Hagan A, Arya N, Guckert M, Schadendorf D, Kefford RF, Grob JJ, Hamid O, Amaravadi R, Simeone E, Wilhelm T, Kim KB, Long GV, Martin AM, Mazumdar J, Goodman VL, Trefzer U. Phase II trial (BREAK-2) of the BRAF inhibitor dabrafenib (GSK2118436) in patients with metastatic melanoma. J Clin Oncol. 2013 Sep 10;31(26):3205-11. doi: 10.1200/JCO.2013.49.8691. Epub 2013 Aug 5. PMID 23918947
- [Derived] Hauschild A, Ascierto PA, Schadendorf D, Grob JJ, Ribas A, Kiecker F, Dutriaux C, Demidov LV, Lebbe C, Rutkowski P, Blank CU, Gutzmer R, Millward M, Kefford R, Haas T, D'Amelio A Jr, Gasal E, Mookerjee B, Chapman PB. Long-term outcomes in patients with BRAF V600-mutant metastatic melanoma receiving dabrafenib monotherapy: Analysis from phase 2 and 3 clinical trials. Eur J Cancer. 2020 Jan;125:114-120. doi: 10.1016/j.ejca.2019.10.033. PMID 31864178
- [Derived] Santiago-Walker A, Gagnon R, Mazumdar J, Casey M, Long GV, Schadendorf D, Flaherty K, Kefford R, Hauschild A, Hwu P, Haney P, O'Hagan A, Carver J, Goodman V, Legos J, Martin AM. Correlation of BRAF Mutation Status in Circulating-Free DNA and Tumor and Association with Clinical Outcome across Four BRAFi and MEKi Clinical Trials. Clin Cancer Res. 2016 Feb 1;22(3):567-74. doi: 10.1158/1078-0432.CCR-15-0321. Epub 2015 Oct 7. PMID 26446943
- [Derived] Ouellet D, Gibiansky E, Leonowens C, O'Hagan A, Haney P, Switzky J, Goodman VL. Population pharmacokinetics of dabrafenib, a BRAF inhibitor: effect of dose, time, covariates, and relationship with its metabolites. J Clin Pharmacol. 2014 Jun;54(6):696-706. doi: 10.1002/jcph.263. Epub 2014 Jan 17. PMID 24408395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants received Dabrafenib (GSK2118436) 150 milligram (mg) twice daily and continued on treatment until disease progression, death, unacceptable adverse event (AE), or early termination of the study. The total duration of the study including a long-term follow-up phase was 5 years.
Pre-assignment Details: A total of 211 participants with histologically confirmed BRAF mutation positive metastatic melanoma (Stage IV) were screened for eligibility. 152 participants had a BRAF V600E or V600K mutation and 92 participants with positive mutation were included in the study.
Groups:
- GSK2118436 150 mg: Participants received GSK2118436 (gelatin capsules) 150 mg orally twice a day and continued on treatment until disease progression, death, or unacceptable AEs . Participants who are benefiting from GSK2118436 at the time of study completion will have the option to enter Study BRF114144 (NCT01231594), which is a rollover study for GSK2118436.
Period: Overall Study
Arm/Group | GSK2118436 150 mg
Started | 92
Completed | 71
Not Completed | 21
Not completed — Study Closed | 16
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (14.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 49
Race/Ethnicity, Customized [Number; unit: participants]
  White | 91
  American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Best Overall Response of Confirmed Complete Response (CR) or Partial Response (PR) as Assessed by the Investigator for Participants Who Had a BRAF V600E Mutation
Description: A participant was defined as a responder if he/she achieved either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter (mm) in the short axis.) or PR (at least a 30 percent decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). To be assigned a status of PR or CR, a confirmatory disease assessment was required at Week 12 if an initial response was seen at the Week 6 scan. Initial responses (CR/PR) that occured at Week 12 or later were required to be confirmed not less than 4 weeks and not more than 6 weeks after the criteria for response were first met. The analysis was performed on Primary efficacy Population which comprised of all participants who received at least one dose of GSK2118436 (All Treated Participants Population) and had a BRAF V600E mutation.
Time Frame: Up to 60 months
Population: Primary efficacy Population
Measure: Number; unit: Participants
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 76
Participants
  CR | 5
  PR | 40
Statistical Analysis 1: Comparison: GSK2118436 150 mg; Test type: Other; percentage of participants = 59, 95% CI 2-sided [48.2 to 70.3] — The estimated value represents the percentage of participants with a confirmed CR or a confirmed PR

2. Secondary Outcome: Number of Participants With a Best Overall Response of CR or PR as Assessed by the Investigator and an Independent Reviewer for Participants Who Had a BRAF V600K Mutation
Description: A participant was defined as a responder if he/she achieved either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or PR (at least a 30 percent decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). To be assigned a status of PR or CR, a confirmatory disease assessment had to have been performed at Week 12 if an initial response was seen at the Week 6 scan. Initial responses (CR/PR) that occured at Week 12 or later should have been confirmed not less than 4 weeks and not more than 6 weeks after the criteria for response were first met. The analysis was performed on Secondary efficacy analysis Population which comprised of all participants who received at least one dose of GSK2118436 (All Treated Participants Population) and had a BRAF V600K mutation.
Time Frame: Up to 60 months
Population: Secondary Efficacy Population
Measure: Number; unit: Participants
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 16
Participants
  Investigator-assessed CR | 0
  Investigator-assessed PR | 2
Statistical Analysis 1: Comparison: GSK2118436 150 mg; Test type: Other; percentage of participants = 13, 95% CI 2-sided [0.0 to 28.7] — The estimated value represents the percentage of participants with a investigator assessed CR or PR

3. Secondary Outcome: Progression-free Survival (PFS) as Assessed by the Investigator and an Independent Reviewer for Participants Who Had a BRAF V600E Mutation
Description: PFS is defined as the interval between the first dose of study medication and the earliest date of disease progression or death due to any cause. The length of this interval is estimated as the date of death or progression minus date of first dose plus 1 day. Kaplan-Meier model was used to estimate the median and 95 percent confidence interval (CI). For participants who received subsequent anti-cancer therapy prior to the date of documented progression or death, PFS was censored at the last adequate assessment. For participants who did not have a documented date of progression or death, PFS was censored at the date of last adequate assessment.
Time Frame: Up to 60 months
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 76
Weeks | 6.3 [4.6 to 8.1]

4. Secondary Outcome: Progression-free Survival (PFS) as Assessed by the Investigator and an Independent Reviewer for Participants Who Had a BRAF V600K Mutation
Description: PFS is defined as the interval between the first dose of study medication and the earliest date of disease progression or death due to any cause. The length of this interval is estimated as the date of death or progression minus date of first dose plus 1 day. Kaplan-Meier model was used to estimate the median and 95 percent CI. For participants who received subsequent anti-cancer therapy prior to the date of documented progression or death, PFS was censored at the last adequate assessment. For participants who did not have a documented date of progression or death, PFS was censored at the date of last adequate assessment.
Time Frame: Up to 60 months
Population: Secondary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 16
Weeks | 4.0 [2.6 to 6.2]

5. Secondary Outcome: Duration of Response as Assessed by the Investigator and an Independent Reviewer for Participants Who Had a BRAF V600E Mutation
Description: Duration of response for participants with either a CR or PR is defined as the time from the first documented evidence of a PR or CR until the first documented sign of disease progression or death due to any cause. Duration of response was estimated using Kaplan-Meier model and the median and 95 percent CI was presented. The analysis was performed on Primary efficacy Population and only those participants who had a CR or PR were analyzed.
Time Frame: Up to 60 months
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 45
Weeks | 6.6 [3.9 to 11.1]

6. Secondary Outcome: Duration of Response as Assessed by the Investigator and an Independent Reviewer for Participants Who Had a BRAF V600K Mutation
Description: Duration of response for participants with either a CR or PR is defined as the time from the first documented evidence of a PR or CR until the first documented sign of disease progression or death due to any cause. Duration of response was estimated using Kaplan-Meier model and the median and 95 percent CI was presented. The analysis was performed on Secondary efficacy Population and only those participants who had a CR or PR were analyzed.
Time Frame: Up to 60 months
Population: Secondary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 3
Weeks | 5.6 [3.7 to 6.8]

7. Secondary Outcome: Overall Survival for Participants Who Had a BRAF V600E Mutation
Description: Overall survival is defined as the time from the first dose of study medication until death due to any cause. For participants who did not die, overall survival was censored at the date of last contact. Overall survival was estimated using kaplan-Meier model and median and 95 percent CI was presented.
Time Frame: Up to 60 months
Population: Primary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 76
Weeks | 13.1 [9.5 to 21.9]
Statistical Analysis 1: Comparison: GSK2118436 150 mg; Test type: Other; percentage of participants = 20, 95% CI 2-sided [11.6 to 29.8] — The estimated value represents the percentage of participants with overall survival

8. Secondary Outcome: Overall Survival for Participants Who Had a BRAF V600K Mutation
Description: as for outcome 7
Time Frame: From the first dose to death due to any cause (up to 60 months)
Population: Secondary Efficacy Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 16
Weeks | 12.9 [4.2 to 17.1]
Statistical Analysis 1: Comparison: GSK2118436 150 mg; Test type: Other; percentage of participants = 13, 95% CI 2-sided [2.2 to 34.6] — The estimated value represents the percentage of participants with overall survival

9. Secondary Outcome: Number of Participants With AEs and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs including systemic allergic and non-allergic reactions as well as local site injection-related reactions were counted throughout treatment phase and follow up phase. Systemic allergic reactions included facial paralysis, flushing, hypersensitivity and rash pruritic. Injection related reactions were considered as systemic non-allergic reactions. Local site reactions included injection site bruising, erythema, pain and reaction. The analysis was performed on All treated Population which comprised of all participants that receive at least one dose of dabrafenib.
Time Frame: Up to 60 months
Population: All treated Population
Measure: Number; unit: Participants
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 92
Participants
  Any AE | 87
  Any SAE | 33

10. Secondary Outcome: Number of Participants With Change From Baseline in Clinical Chemistry and Hematology Toxicity Grades
Description: Blood samples were collected from participants for evaluation of change from Baseline in toxicity grades in clinical chemistry and hematology parameters. The clinical chemistry parameters included alkaline phosphatase, Alanine amino transferase (ALT), Aspartate amino transferase (AST), total bilirubin, creatinine, glucose, potassium, magnesium, sodium and phosphorus. The hematology parameters included hemoglobin, total neutrophils, platelets and white blood cells (WBC). Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. The change from Baseline was calculated as visit value minus Baseline value and was presented in the form of worst case post-baseline value which was the maximum toxicity grade for a participant after the first dose of study drug over the treatment period. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Up to 60 months
Population: All treated Population
Measure: Number; unit: Participants
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 92
Participants
  Alkaline phosphatase; n= 91: number analyzed (Participants) | 91
  Alkaline phosphatase; n= 91 | 23
  ALT; n= 91: number analyzed (Participants) | 91
  ALT; n= 91 | 18
  AST; n= 91: number analyzed (Participants) | 91
  AST; n= 91 | 18
  Total bilirubin; n= 91: number analyzed (Participants) | 91
  Total bilirubin; n= 91 | 3
  Creatinine; n= 91: number analyzed (Participants) | 91
  Creatinine; n= 91 | 11
  Glucose; n= 90: number analyzed (Participants) | 90
  Glucose; n= 90 | 51
  Potassium; n= 91: number analyzed (Participants) | 91
  Potassium; n= 91 | 2
  Magnesium; n= 89: number analyzed (Participants) | 89
  Magnesium; n= 89 | 2
  Sodium; n= 91: number analyzed (Participants) | 91
  Sodium; n= 91 | 5
  Phosphorus; n= 91: number analyzed (Participants) | 91
  Phosphorus; n= 91 | 36
  Hemoglobin; n= 91: number analyzed (Participants) | 91
  Hemoglobin; n= 91 | 0
  Total Neutrophils; n= 91: number analyzed (Participants) | 91
  Total Neutrophils; n= 91 | 21
  Platelet; n= 91: number analyzed (Participants) | 91
  Platelet; n= 91 | 12
  WBC; n= 91: number analyzed (Participants) | 91
  WBC; n= 91 | 24

11. Secondary Outcome: Number of Participants With Change From Baseline in Temperature and Pulse Rate
Description: Number of participants with change from Baseline in temperature and pulse rate were evaluated from the first dose of study treatment till discontinuation due to any reason. Change from Baseline in worst-case post Baseline value was presented as decrease to <=35, change to normal or no change and increase to >=38. Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. The change from Baseline was calculated as visit value minus Baseline value and was presented in the form of worst case post-baseline value which was the maximum toxicity grade for a participant after the first dose of study drug over the treatment period.
Time Frame: Up to 60 months
Population: All treated Population
Measure: Number; unit: Participants
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 91
Participants
  Temperature; Decrease to <=35 | 3
  Temperature; Change to normal or no change | 84
  Temperature; Increase to >=38 | 4
  Pulse rate; Decrease to <=35 | 9
  Pulse rate; Change to normal or no change | 66
  Pulse rate; Increase to >=38 | 16

12. Secondary Outcome: Number of Participants With Increase From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Number of participants with increase from Baseline in SBP and DBP were evaluated from the first dose of study treatment till discontinuation due to any reason. Change from Baseline in worst-case post Baseline value was presented as any increase to >=80 and increase to >=100 for DBP and as any increase to >=120 and increase to >=160 for SBP. Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. The change from Baseline was calculated as visit value minus Baseline value and was presented in the form of worst-case post Baseline value which was the maximum toxicity grade for a participant after the first dose of study drug over the treatment period. One participant out of the 92 participants (76 BRAF V600E patients + 16 BRAF V600K patients) did not have SBP and DBP collected after baseline.
Time Frame: Up to 60 months
Population: All treated Population
Measure: Number; unit: Participants
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 91
Participants
  DBP; Any increase to >=80 | 32
  DBP; Increase to >=100 | 6
  SBP; Any icrease to >=120 | 2
  SBP; Increase to >=160 | 7

13. Secondary Outcome: Number of Participants With Change From Baseline in Left Ventricular Ejection Fraction (LVEF) Levels
Description: LVEF was defined as the percentage of blood pumped out of the left ventricle. Change from Baseline in worst-case post Baseline was presented as no change or any increase and any decrease values. Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. The change from Baseline was calculated as visit value minus Baseline value and was presented in the form of worst-case post Baseline value which was the maximum toxicity grade for a participant after the first dose of study drug over the treatment period.
Time Frame: Up to 60 months
Population: All treated Population
Measure: Number; unit: Participants
Arm/Group | GSK2118436 150 mg
Number analyzed (Participants) | 92
Participants
  No change or any increase | 34
  Any decrease | 54

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of investigational product until death of all participants or a follow-up till 60 months.
Description: SAEs and non-serious AEs were collected in the All Treated Participants Population, comprised of all randomized participants who received at least one dose of study medication, according to the actual treatment received.
Arm/Group | GSK2118436 150 mg
All-Cause Mortality (participants affected / at risk) | 71/92
Serious Adverse Events (participants affected / at risk) | 33/92
Other Adverse Events (participants affected / at risk) | 83/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2118436 150 mg (N=92)
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Arrhythmia supraventricular (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Adverse drug reaction (General disorders) | 1
Chills (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pyrexia (General disorders) | 4
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Post procedural hematoma (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Aphasia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Miscarriage of partner (Social circumstances) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2118436 150 mg (N=92)
Anaemia (Blood and lymphatic system disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 7
Tachycardia (Cardiac disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 8
Chills (General disorders) | 13
Fatigue (General disorders) | 22
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 24
Bronchitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 13
Blood alkaline phosphatase increased (Investigations) | 5
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 33
Back pain (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15
Headache (Nervous system disorders) | 19
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Actinic keratosis (Skin and subcutaneous tissue disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 11
Erythema (Skin and subcutaneous tissue disorders) | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 27
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 9
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 10
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 6
Hot flush (Vascular disorders) | 6

LIMITATIONS AND CAVEATS:
This study met the criteria for completed. Participants who were still receiving study treatment at the time the study was closed were given the option to transfer to a rollover protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.